CLINICAL TRIAL: NCT02648204
Title: Efficacy and Safety of Semaglutide Versus Dulaglutide as add-on to Metformin in Subjects With Type 2 Diabetes
Acronym: SUSTAIN 7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4216; 2014-005375-91 (EudraCT Number); U1111-1164-8495 (Other: WHO)
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Semaglutide 0.5 mg/Week (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide 1.0 mg/Week (Experimental)
  Interventions: Drug: semaglutide
- Dulaglutide 0.75 mg/Week (Active Comparator)
  Interventions: Drug: Dulaglutide
- Dulaglutide 1.5 mg/Week (Active Comparator)
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: semaglutide — Administered subcutaneously (s.c., under the skin) once-weekly.
  Arms: Semaglutide 0.5 mg/Week; Semaglutide 1.0 mg/Week
Drug: Dulaglutide — Administered subcutaneously (s.c., under the skin) once-weekly.
  Arms: Dulaglutide 0.75 mg/Week; Dulaglutide 1.5 mg/Week

SUMMARY:
This trial is conducted in Asia, Europe and the United States of America (USA). The aim of the trial is to investigate efficacy and safety of semaglutide versus dulaglutide as add-on to metformin in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Male or female, age at least 18 years at the time of signing informed consent. - HbA1c (glycosylated haemoglobin) 7.0 - 10.5% (53 - 91 mmol/mol) (both inclusive) - Subjects on stable diabetes treatment with metformin (minimum of 1500 mg/day or maximal tolerated dose documented in the patient medical record) for 90 days prior to screening Exclusion Criteria: - Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice) - Any condition, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol - Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before screening. An exception is short-term insulin treatment for acute illness for a total of equal to or below 14 days - History of pancreatitis (acute or chronic) - Screening calcitonin equal to or above 50 ng/L - Family or personal history of Multiple Endocrine Neoplasia Type 2 or Medullary Thyroid Carcinoma - Renal impairment defined as eGFR (electronic case report form) below 60 mL/min/1.73 m^2 as per CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) - Subjects presently classified as being in New York Heart Association Class IV - Planned coronary, carotid or peripheral artery revascularisation on the day of screening - Proliferative retinopathy or maculopathy requiring acute treatment - History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and in-situ carcinomas) - Anticipated initiation or change in concomitant medications (for more than 14 consecutive days or on a frequent basis) known to affect weight or glucose metabolism (e.g. orlistat, thyroid hormones, corticosteroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1201 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (180):
- United States (88):
  - Novo Nordisk Investigational Site, Tuscumbia, Alabama
  - Novo Nordisk Investigational Site, Chandler, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Buena Park, California
  - Novo Nordisk Investigational Site, Carlsbad, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Huntington Park, California
  - Novo Nordisk Investigational Site, Lincoln, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Riverside, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Van Nuys, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Norwalk, Connecticut
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Coral Gables, Florida
  - Novo Nordisk Investigational Site, Edgewater, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Port Orange, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Adairsville, Georgia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Bainbridge, Georgia
  - Novo Nordisk Investigational Site, Conyers, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Suwanee, Georgia
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Addison, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Gillespie, Illinois
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Greenfield, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Newton, Kansas
  - Novo Nordisk Investigational Site, Park City, Kansas
  - Novo Nordisk Investigational Site, Covington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Owensboro, Kentucky
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Oxon Hill, Maryland
  - Novo Nordisk Investigational Site, Methuen, Massachusetts
  - Novo Nordisk Investigational Site, Rochester, Michigan
  - Novo Nordisk Investigational Site, Port Gibson, Mississippi
  - Novo Nordisk Investigational Site, Missoula, Montana
  - Novo Nordisk Investigational Site, Trenton, New Jersey
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Garner, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Wadsworth, Ohio
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Corvallis, Oregon
  - Novo Nordisk Investigational Site, Fleetwood, Pennsylvania
  - Novo Nordisk Investigational Site, Harleysville, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Moncks Corner, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Rapid City, South Dakota
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Katy, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Riverton, Utah
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Walla Walla, Washington
  - Novo Nordisk Investigational Site, Wenatchee, Washington
- Bulgaria (5):
  - Novo Nordisk Investigational Site, Blagoevgrad
  - Novo Nordisk Investigational Site, Burgas
  - Novo Nordisk Investigational Site, Montana
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Stara Zagora
- Croatia (6):
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Krapinske Toplice
  - Novo Nordisk Investigational Site, Rijeka
  - Novo Nordisk Investigational Site, Varaždin
  - Novo Nordisk Investigational Site, Virovitica
  - Novo Nordisk Investigational Site, Zagreb
- Finland (6):
  - Novo Nordisk Investigational Site, Jyväskylä
  - Novo Nordisk Investigational Site, Kerava
  - Novo Nordisk Investigational Site, Kuusamo
  - Novo Nordisk Investigational Site, Raisio
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- Germany (7):
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
- Greece (5):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Chalkida, Evia
  - Novo Nordisk Investigational Site, Ioannina
  - Novo Nordisk Investigational Site, Piraeus
  - Novo Nordisk Investigational Site, Thessaloniki
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- India (22):
  - Novo Nordisk Investigational Site, Guntur, Andhra Pradesh
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Visakhapatnam, Andhra Pradesh
  - Novo Nordisk Investigational Site, Guwahati, Assam
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Kozhikode, Kerala
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Goa, Maharashtra
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Delhi, New Delhi
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Bhubaneswar, Odisha
  - Novo Nordisk Investigational Site, Mohali, Punjab
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, Ludhiana
  - Novo Nordisk Investigational Site, New Delhi
- Ireland (3):
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Galway
  - Novo Nordisk Investigational Site, Gorey
- Novo Nordisk Investigational Site, Riga, Latvia
- Lithuania (3):
  - Novo Nordisk Investigational Site, Kaunas
  - Novo Nordisk Investigational Site, Panevezys
  - Novo Nordisk Investigational Site, Vilnius
- Portugal (6):
  - Novo Nordisk Investigational Site, Almada
  - Novo Nordisk Investigational Site, Aveiro
  - Novo Nordisk Investigational Site, Lisbon
  - Novo Nordisk Investigational Site, Tomar
  - Novo Nordisk Investigational Site, Viana do Castelo
  - Novo Nordisk Investigational Site, Vila Nova de Gaia
- Novo Nordisk Investigational Site, Ponce, Puerto Rico
- Romania (6):
  - Novo Nordisk Investigational Site, Oradea, Bihor County
  - Novo Nordisk Investigational Site, Târgu Mureş, Mureș County
  - Novo Nordisk Investigational Site, Brasov
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Buzău
  - Novo Nordisk Investigational Site, Galati
- Slovakia (5):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Levice
  - Novo Nordisk Investigational Site, Piešťany
  - Novo Nordisk Investigational Site, Poprad
  - Novo Nordisk Investigational Site, Prievidza
- Spain (8):
  - Novo Nordisk Investigational Site, Alicante
  - Novo Nordisk Investigational Site, La Roca Del Vallés
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Segovia
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Vic (Barcelona)
- United Kingdom (7):
  - Novo Nordisk Investigational Site, Bradford-on-Avon
  - Novo Nordisk Investigational Site, Northwood
  - Novo Nordisk Investigational Site, Romford
  - Novo Nordisk Investigational Site, Soham
  - Novo Nordisk Investigational Site, Southampton
  - Novo Nordisk Investigational Site, Stevenage
  - Novo Nordisk Investigational Site, Watford

REFERENCES:
- [Background] Rodbard HW, Bellary S, Hramiak I, Seino Y, Silver R, Damgaard LH, Nayak G, Zacho J, Aroda VR. GREATER COMBINED REDUCTIONS IN HbA1C >/=1.0% AND WEIGHT >/=5.0% WITH SEMAGLUTIDE VERSUS COMPARATORS IN TYPE 2 DIABETES. Endocr Pract. 2019 Jun;25(6):589-597. doi: 10.4158/EP-2018-0444. Epub 2019 Mar 13. PMID 30865526
- [Background] Johansen P, Hakan-Bloch J, Liu AR, Bech PG, Persson S, Leiter LA. Cost Effectiveness of Once-Weekly Semaglutide Versus Once-Weekly Dulaglutide in the Treatment of Type 2 Diabetes in Canada. Pharmacoecon Open. 2019 Dec;3(4):537-550. doi: 10.1007/s41669-019-0131-6. PMID 30927241
- [Background] Malkin SJP, Russel-Szymczyk M, Psota M, Hlavinkova L, Hunt B. The Management of Type 2 Diabetes with Once-Weekly Semaglutide Versus Dulaglutide: A Long-Term Cost-Effectiveness Analysis in Slovakia. Adv Ther. 2019 Aug;36(8):2034-2051. doi: 10.1007/s12325-019-00965-y. Epub 2019 Jun 5. PMID 31168765
- [Result] Pratley RE, Aroda VR, Lingvay I, Ludemann J, Andreassen C, Navarria A, Viljoen A; SUSTAIN 7 investigators. Semaglutide versus dulaglutide once weekly in patients with type 2 diabetes (SUSTAIN 7): a randomised, open-label, phase 3b trial. Lancet Diabetes Endocrinol. 2018 Apr;6(4):275-286. doi: 10.1016/S2213-8587(18)30024-X. Epub 2018 Feb 1. PMID 29397376
- [Result] Ahmann AJ, Capehorn M, Charpentier G, Dotta F, Henkel E, Lingvay I, Holst AG, Annett MP, Aroda VR. Efficacy and Safety of Once-Weekly Semaglutide Versus Exenatide ER in Subjects With Type 2 Diabetes (SUSTAIN 3): A 56-Week, Open-Label, Randomized Clinical Trial. Diabetes Care. 2018 Feb;41(2):258-266. doi: 10.2337/dc17-0417. Epub 2017 Dec 15. PMID 29246950
- [Result] Sharma R, Wilkinson L, Vrazic H, Popoff E, Lopes S, Kanters S, Druyts E. Comparative efficacy of once-weekly semaglutide and SGLT-2 inhibitors in type 2 diabetic patients inadequately controlled with metformin monotherapy: a systematic literature review and network meta-analysis. Curr Med Res Opin. 2018 Sep;34(9):1595-1603. doi: 10.1080/03007995.2018.1476332. Epub 2018 May 29. PMID 29764222
- [Result] Wilkinson L, Hunt B, Johansen P, Iyer NN, Dang-Tan T, Pollock RF. Cost of Achieving HbA1c Treatment Targets and Weight Loss Responses with Once-Weekly Semaglutide Versus Dulaglutide in the United States. Diabetes Ther. 2018 Jun;9(3):951-961. doi: 10.1007/s13300-018-0402-8. Epub 2018 Mar 19. PMID 29557057
- [Result] Aroda VR, Ahmann A, Cariou B, Chow F, Davies MJ, Jodar E, Mehta R, Woo V, Lingvay I. Comparative efficacy, safety, and cardiovascular outcomes with once-weekly subcutaneous semaglutide in the treatment of type 2 diabetes: Insights from the SUSTAIN 1-7 trials. Diabetes Metab. 2019 Oct;45(5):409-418. doi: 10.1016/j.diabet.2018.12.001. Epub 2019 Jan 4. PMID 30615985
- [Result] Viljoen A, Hoxer CS, Johansen P, Malkin S, Hunt B, Bain SC. Evaluation of the long-term cost-effectiveness of once-weekly semaglutide versus dulaglutide for treatment of type 2 diabetes mellitus in the UK. Diabetes Obes Metab. 2019 Mar;21(3):611-621. doi: 10.1111/dom.13564. Epub 2018 Nov 28. PMID 30362224
- [Derived] Osumili B, Fan L, Paik JS, Pantalone KM, Ranta K, Sapin H, Tofe S. Tirzepatide 5, 10 and 15 mg versus injectable semaglutide 0.5 mg for the treatment of type 2 diabetes: An adjusted indirect treatment comparison. Diabetes Res Clin Pract. 2024 Jun;212:111717. doi: 10.1016/j.diabres.2024.111717. Epub 2024 May 21. PMID 38777128
- [Derived] Pratley RE, Aroda VR, Catarig AM, Lingvay I, Ludemann J, Yildirim E, Viljoen A. Impact of patient characteristics on efficacy and safety of once-weekly semaglutide versus dulaglutide: SUSTAIN 7 post hoc analyses. BMJ Open. 2020 Nov 16;10(11):e037883. doi: 10.1136/bmjopen-2020-037883. PMID 33199417
- [Derived] DeSouza C, Cariou B, Garg S, Lausvig N, Navarria A, Fonseca V. Efficacy and Safety of Semaglutide for Type 2 Diabetes by Race and Ethnicity: A Post Hoc Analysis of the SUSTAIN Trials. J Clin Endocrinol Metab. 2020 Feb 1;105(2):dgz072. doi: 10.1210/clinem/dgz072. PMID 31769496
- [Derived] Jendle J, Birkenfeld AL, Polonsky WH, Silver R, Uusinarkaus K, Hansen T, Hakan-Bloch J, Tadayon S, Davies MJ. Improved treatment satisfaction in patients with type 2 diabetes treated with once-weekly semaglutide in the SUSTAIN trials. Diabetes Obes Metab. 2019 Oct;21(10):2315-2326. doi: 10.1111/dom.13816. Epub 2019 Jul 12. PMID 31215727
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 210 sites were approved for recruiting subjects, of which 196 sites randomized the subjects: Bulgaria: 6; Croatia: 6; Finland: 6; Germany: 6; Greece: 8; Hong Kong: 1; India: 22; Ireland: 5; Latvia: 3; Lithuania: 5; Portugal: 4; Romania: 7; Slovakia: 6; Spain: 8; United Kingdom: 8; United States: 95.
Groups:
- Semaglutide 0.5 mg: Subjects received subcutaneous (s.c., under the skin) injections of semaglutide once weekly (OW) for treatment duration of 40 weeks. Subjects received semaglutide 0.25 mg for 4 weeks (weeks 1 to 4) followed by 0.5 mg for 36 weeks (weeks 5 to 40).
- Semaglutide 1.0 mg: Subjects received s.c. injections of semaglutide OW for treatment duration of 40 weeks. Subjects received semaglutide 0.25 mg for 4 weeks (week 1 to 4) followed by 0.5 mg for another 4 weeks (week 5 to 8) and then semaglutide 1.0 mg for remaining 32 weeks (week 9-40). Subjects were followed for 5 weeks after completion of treatment period.
- Dulaglutide 0.75 mg: Subjects received s.c. injections of dulaglutide 0.75 mg OW for treatment duration of 40 weeks. Subjects were followed for 5 weeks after completion of treatment period.
- Dulaglutide 1.5 mg: Subjects received s.c. injections of dulaglutide 1.5 mg OW for treatment duration of 40 weeks. Subjects were followed for 5 weeks after completion of treatment period.
Period: Overall Study
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Started | 301 | 300 | 300 | 300
Exposed | 301 | 300 | 299 | 299
Completed | 279 | 279 | 287 | 284
Not Completed | 22 | 21 | 13 | 16
Not completed — Withdrawal by Subject | 12 | 8 | 2 | 6
Not completed — Lost to Follow-up | 5 | 8 | 4 | 6
Not completed — Missing follow-up information | 4 | 4 | 4 | 2
Not completed — Death | 1 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised subjects exposed to at least one dose of trial product. Subjects in the FAS would contribute to the evaluation "as randomised".
Groups:
- Semaglutide 0.5 mg: Subjects received s.c. injections of semaglutide OW for treatment duration of 40 weeks. Subjects received semaglutide 0.25 mg for 4 weeks (weeks 1 to 4) followed by 0.5 mg for 36 weeks (weeks 5 to 40).
- Semaglutide 1.0 mg: Subjects received s.c. injections of semaglutide OW for treatment duration of 40 weeks. Subjects received semaglutide 0.25 mg for 4 weeks (weeks 1 to 4) followed by 0.5 mg for another 4 weeks (weeks 5 to 8) and then semaglutide 1.0 mg for remaining 32 weeks (weeks 9-40). Subjects were followed for 5 weeks after completion of treatment period.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg | Total
Number analyzed (Participants) | 301 | 300 | 299 | 299 | 1199
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (10.9) | 55 (10.6) | 55 (10.4) | 56 (10.6) | 56 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 162 | 160 | 171 | 662
  Male | 132 | 138 | 139 | 128 | 537
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 35 | 31 | 43 | 138
  Not Hispanic or Latino | 272 | 265 | 268 | 256 | 1061
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 50 | 38 | 48 | 55 | 191
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 17 | 18 | 17 | 18 | 70
  White | 233 | 243 | 232 | 220 | 928
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 6 | 10
Glycosylated haemoglobin (Hb1Ac) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.3 (0.96) | 8.2 (0.92) | 8.2 (0.91) | 8.2 (0.89) | 8.2 (0.92)
Body weight [Mean (Standard Deviation); unit: kg] | 96.4 (24.38) | 95.5 (20.90) | 95.6 (23.01) | 93.4 (21.79) | 95.2 (22.56)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] — Population: Number of subjects analysed=subjects with available data of fasting plasma glucose at baseline
  mmol/L
    number analyzed (Participants) | 298 | 299 | 297 | 297 | 1191
    (all) | 9.8 (2.54) | 9.8 (2.58) | 9.7 (2.65) | 9.6 (2.29) | 9.7 (2.52)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Results are based on HbA1c data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on-treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. The post-baseline responses are analysed using a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: Week 0, week 40
Population: Analysis was based on FAS.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 299
percentage of HbA1c | -1.51 (0.06) | -1.78 (0.06) | -1.11 (0.05) | -1.37 (0.06)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Dulaglutide 0.75 mg; Test type: Non-Inferiority — Non-Inferiority margin: 0.4; p < 0.0001, Mixed Models Analysis; Treatment difference = -0.40, 95% CI 2-sided [-0.55 to -0.25], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Semaglutide 0.5 mg vs Dulaglutide 0.75 mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Treatment difference = -0.40, 95% CI 2-sided [-0.55 to -0.25], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Semaglutide 1.0 mg vs Dulaglutide 1.5 mg; Test type: Non-Inferiority — Non-Inferiority margin: 0.04; p < 0.0001, Mixed Models Analysis; Treatment difference = -0.41, 95% CI 2-sided [-0.57 to -0.25], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Semaglutide 1.0 mg vs Dulaglutide 1.5 mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Treatment difference = -0.41, 95% CI 2-sided [-0.57 to -0.25], Standard Error of Mean 0.08

2. Secondary Outcome: Change in Body Weight (kg)
Description: Results are based on body weight data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication.
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of subjects analysed=number of subjects with available data for body weight.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 298
kg | -4.56 (0.28) | -6.53 (0.28) | -2.30 (0.27) | -2.98 (0.27)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Dulaglutide 0.75 mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Treatment difference = -2.26, 95% CI 2-sided [-3.02 to -1.51], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Dulaglutide 1.5 mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Treatment difference = -3.55, 95% CI 2-sided [-4.32 to -2.78], Standard Error of Mean 0.39

3. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Results are based on fasting plasma glucose data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication.
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for fasting plasma glucose.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 298 | 299 | 297 | 297
mmol/L | -2.18 (0.12) | -2.83 (0.12) | -1.87 (0.12) | -2.25 (0.12)

4. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: Results are based on systolic and diastolic blood pressure data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication.
Time Frame: Week 0, week 40
Population: Analysis was based on FAS.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 299
mmHg
  Diastolic BP | -0.57 (0.48) | -2.05 (0.49) | -0.35 (0.47) | -0.03 (0.47)
  Systolic BP | -2.44 (0.76) | -4.88 (0.77) | -2.16 (0.75) | -2.86 (0.75)

5. Secondary Outcome: Change in Overall Scores for Patient Reported Outcomes: Diabetes Treatment Satisfaction Questionnaire
Description: The questionnaire contains 8 items and evaluates subjects' diabetes treatment in terms of convenience, flexibility and general feelings towards treatment. The result presented is 'Treatment Satisfaction' summary score (sum of 6 of the 8 items). Response options: 6 (best case) to 0 (worst case). Total scores range: 0-36. Higher scores=higher satisfaction. Results are based on data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was period where subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This includes observations recorded at, or after the date of first dose of trial product and not after first occurrence of following: the end-date of the 'on-treatment' observation period or initiation of rescue medication
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for diabetes treatment satisfaction questionnaire
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 299 | 299 | 298
units on a scale | 4.60 (0.28) | 4.55 (0.29) | 4.52 (0.28) | 4.65 (0.28)

6. Secondary Outcome: HbA1c Below or Equal to 6.5% (48 mmol/Mol) American Association of Clinical Endocrinologists Target
Description: Percentage of subjects who achieved HbA1c target below or equal to 6.5% (48 mmol/mol) after 40 weeks of treatment. Results are based on data from on-treatment without rescue medication period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. Missing data imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: After 40 weeks treatment
Population: Results are based on the FAS.
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 299
percentage of subjects
  Yes | 49.2 | 66.7 | 34.1 | 47.2
  No | 50.8 | 33.3 | 65.9 | 52.8

7. Secondary Outcome: Change From Baseline in 7-point Self-measured Plasma Glucose (SMPG) Mean Profile
Description: SMPG values were recorded at 7 time-points: before and 90 minutes after start of breakfast, lunch, and dinner, and at bedtime. Reported results are mean profile from on-treatment without rescue medication observation period. The 'on-treatment' observation period was period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. The post-baseline responses are analysed using a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of participants analysed=Number of participants analysed=number of participants with available data for 7-point self-measured plasma glucose.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 295 | 295 | 296 | 296
mmol/L | -2.43 (0.10) | -2.95 (0.10) | -1.99 (0.10) | -2.32 (0.10)

8. Secondary Outcome: Change From Baseline 7-point Self-measured Plasma Glucose Increment
Description: SMPG values were recorded at 7 time-points: before and 90 minutes after start of breakfast, lunch, and dinner, and at bedtime. Reported results are plasma glucose incremental profile from on-treatment without rescue medication observation period. The 'on-treatment' observation period was period where subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes observations recorded at, or after date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. The post-baseline responses are analysed using a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for 7-point self-measured plasma glucose increment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 295 | 292 | 296 | 296
mmol/L | -0.77 (0.08) | -0.93 (0.09) | -0.44 (0.08) | -0.63 (0.08)

9. Secondary Outcome: Change in Fasting Blood Lipids (Total Cholesterol)
Description: Results are based on the data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. The post-baseline responses are analysed using a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit. Change from baseline is presented in terms of ratio to baseline value.
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for total cholesterol
Measure: Geometric Least Squares Mean (Standard Error); unit: ratio to baseline
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 295 | 296 | 290 | 294
ratio to baseline | 0.96 (0.01) | 0.97 (0.01) | 0.97 (0.01) | 0.99 (0.01)

10. Secondary Outcome: Change in Fasting Blood Lipids (Low Density Lipoprotein [LDL] Cholesterol)
Description: as for outcome 9
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for LDL cholesterol.
Measure: Geometric Least Squares Mean (Standard Error); unit: ratio to baseline
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 293 | 295 | 290 | 294
ratio to baseline | 0.97 (0.02) | 1.00 (0.02) | 0.97 (0.02) | 1.01 (0.02)

11. Secondary Outcome: Change in Fasting Blood Lipids (High Density Lipoprotein [HDL] Cholesterol)
Description: as for outcome 9
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for HDL cholesterol.
Measure: Geometric Least Squares Mean (Standard Error); unit: ratio to baseline
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 293 | 296 | 290 | 294
ratio to baseline | 0.99 (0.01) | 1.01 (0.01) | 1.00 (0.01) | 1.02 (0.01)

12. Secondary Outcome: Change in Fasting Blood Lipids (Triglycerides)
Description: as for outcome 9
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for triglycerides.
Measure: Geometric Least Squares Mean (Standard Error); unit: ratio to baseline
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 293 | 296 | 290 | 294
ratio to baseline | 0.91 (0.02) | 0.86 (0.02) | 0.91 (0.02) | 0.90 (0.02)

13. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Results are based on the data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. The post-baseline responses are analysed using a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for BMI.
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 298
kg/m^2 | -1.63 (0.10) | -2.33 (0.10) | -0.82 (0.10) | -1.08 (0.10)

14. Secondary Outcome: Change in Waist Circumference
Description: as for outcome 13
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for waist circumference.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 299 | 300 | 298 | 297
cm | -4.27 (0.34) | -5.20 (0.34) | -2.36 (0.33) | -2.93 (0.33)

15. Secondary Outcome: Change in Short Form Health Survey (SF-36v2™)
Description: The questionnaire contains 36 items across 8 domains and 2 summary scores. Score range: 0 (worst score) to 100 (best score). Results are based on the data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was period where subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. The post-baseline responses are analysed using a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: Week 0, week 40
Population: Analysis was based on FAS. Number analysed=number of participants with available data for SF-36.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 299
units on a scale
  Physical component summary: number analyzed (Participants) | 300 | 299 | 295 | 298
  Physical component summary | 1.21 (0.40) | 2.04 (0.40) | 1.93 (0.39) | 1.29 (0.39)
  Mental component summary: number analyzed (Participants) | 300 | 299 | 295 | 298
  Mental component summary | 1.45 (0.49) | 1.23 (0.49) | 0.95 (0.48) | 1.08 (0.48)
  Physical functioning: number analyzed (Participants) | 301 | 300 | 298 | 299
  Physical functioning | 1.25 (0.44) | 2.00 (0.44) | 2.17 (0.43) | 1.05 (0.43)
  Role-physical: number analyzed (Participants) | 300 | 299 | 298 | 299
  Role-physical | 0.98 (0.48) | 2.03 (0.48) | 1.39 (0.47) | 0.82 (0.47)
  Bodily pain: number analyzed (Participants) | 301 | 299 | 299 | 299
  Bodily pain | 0.96 (0.52) | 1.54 (0.52) | 1.69 (0.51) | 0.77 (0.51)
  General health: number analyzed (Participants) | 301 | 299 | 298 | 299
  General health | 2.65 (0.43) | 2.52 (0.43) | 1.86 (0.42) | 2.73 (0.42)
  Vitality: number analyzed (Participants) | 301 | 299 | 299 | 299
  Vitality | 1.23 (0.50) | 1.97 (0.50) | 2.14 (0.49) | 1.83 (0.50)
  Social functioning: number analyzed (Participants) | 301 | 299 | 299 | 299
  Social functioning | 1.18 (0.49) | 0.83 (0.49) | 0.78 (0.48) | 0.63 (0.48)
  Role-emotional: number analyzed (Participants) | 300 | 299 | 297 | 298
  Role-emotional | 1.11 (0.57) | 1.57 (0.58) | 1.04 (0.56) | 1.08 (0.57)
  Mental health: number analyzed (Participants) | 301 | 299 | 299 | 299
  Mental health | 1.89 (0.49) | 1.65 (0.49) | 1.43 (0.48) | 0.96 (0.48)

16. Secondary Outcome: Subjects Who After 40 Weeks Treatment Achieve (Yes/no) HbA1c <7.0% (53 mmol/Mol) American Diabetes Association (ADA) Target
Description: Percentage of subjects who achieved HbA1c target below or equal to <7.0% (53 mmol/mol) after 40 weeks of treatment. Results are based on data from on-treatment without rescue medication period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. Missing data imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: After 40 weeks of treatment
Population: Analysis was based on FAS.
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 299
percentage of subjects
  Yes | 68.4 | 78.7 | 52.2 | 66.6
  No | 31.6 | 21.3 | 47.8 | 33.4

17. Secondary Outcome: Subjects Who After 40 Weeks Treatment Achieve (Yes/no) Weight Loss ≥5%
Description: Percentage of subjects who achieved weight loss ≥5% after 40 weeks of treatment. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. Missing data imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: After 40 weeks treatment
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for body weight.
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 298
percentage of subjects
  Yes | 43.9 | 63.0 | 22.7 | 30.2
  No | 56.1 | 37.0 | 77.3 | 69.8

18. Secondary Outcome: Subjects Who After 40 Weeks Treatment Achieve (Yes/no) Weight Loss ≥10%
Description: Percentage of subjects who achieved weight loss ≥10% after 40 weeks of treatment. Results are based on the data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. Missing data imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: After 40 weeks treatment
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for body weight
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 298
percentage of subjects
  Yes | 14.3 | 26.7 | 3.3 | 7.7
  No | 85.7 | 73.3 | 96.7 | 92.3

19. Secondary Outcome: Subjects Who After 40 Weeks Treatment Achieve (Yes/no) HbA1c <7.0% (53 mmol/Mol) Without Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemia Episodes and no Weight Gain
Description: Percentage of subjects achieved (yes/no) HbA1c <7.0% (53 mmol/mol) without severe or BG confirmed symptomatic hypoglycaemia episodes and no weight gain after 40 weeks of treatment. Results are based on data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was period where subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was subset of 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. Missing data imputed from mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit
Time Frame: After 40 weeks of treatment
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for this endpoint.
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 298
percentage of subjects
  Yes | 64.5 | 74.0 | 44.1 | 58.4
  No | 35.5 | 26.0 | 55.9 | 41.6

20. Secondary Outcome: Subjects Who After 40 Weeks Treatment Achieve (Yes/no) HbA1c Reduction ≥1%
Description: Percentage of subjects who achieved (yes/no) HbA1c reduction of ≥1% after 40 weeks of treatment. Results are based on the data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. Missing data imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: After 40 weeks of treatment
Population: Analysis was based on FAS.
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 299
percentage of subjects
  Yes | 77.4 | 83.3 | 53.8 | 67.6
  No | 22.6 | 16.7 | 46.2 | 32.4

21. Secondary Outcome: Subjects Who After 40 Weeks Treatment Achieve (Yes/no) Weight Loss ≥3%
Description: Percentage of subjects who achieved (yes/no) weight loss of ≥3% after 40 weeks of treatment. Results are based on the data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. Missing data imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: After 40 weeks treatment
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for body weight
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 298
percentage of subjects
  Yes | 64.5 | 76.7 | 36.5 | 44.6
  No | 35.5 | 23.3 | 63.5 | 55.4

22. Secondary Outcome: Subjects Who After 40 Weeks Treatment Achieve (Yes/no) HbA1c Reduction ≥1% and Weight Loss ≥3%
Description: Percentage of subjects who achieved (yes/no) HbA1c reduction ≥1% and weight loss ≥3% 40 weeks of treatment. Results are based on the data from on-treatment without rescue medication observation period. The 'on-treatment' observation period was the period where the subject was considered to be exposed to trial product. The 'on-treatment without rescue medication' observation period was a subset of the 'on -treatment' observation period, where subjects did not receive any non-investigational antidiabetic medication (rescue medication). This period includes the observations recorded at, or after the date of first dose of trial product and not after the first occurrence of the following: the end-date of the 'on-treatment' observation period or initiation of rescue medication. Missing data imputed from a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: After 40 weeks treatment
Population: Analysis was based on FAS. Number of participants analysed=number of participants with available data for HbA1c and body weight.
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 298
percentage of subjects
  Yes | 53.2 | 68.3 | 25.1 | 34.9
  No | 46.8 | 31.7 | 74.9 | 65.1

23. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an AE with onset in the 'on-treatment' period (information collected while subjects were considered as exposed to trial product). This corresponded to information collected until the follow-up (5 weeks after the last treatment including a visit window of +7 days).
Time Frame: 40 weeks + follow-up of 5 weeks
Population: Analysis was based on the safety analysis set which included all randomised subjects exposed to at least one dose of trial product.
Measure: Number; unit: events
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 299
events | 966 | 1015 | 802 | 957

24. Secondary Outcome: Number of Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemia Episodes
Description: A treatment emergent hypoglycaemic episode was defined as an episode with onset in the 'on-treatment' period (information collected while subjects were considered as exposed to trial product). This corresponded to information collected until the follow-up (5 weeks after the last treatment including a visit window of +7 days). Severe or BG-confirmed symptomatic hypoglycaemia was defined as an episode that was severe according to the American Diabetes Association classification or BG-confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: 40 weeks + follow-up of 5 weeks
Population: as for outcome 23
Measure: Number; unit: hypoglycaemic episodes
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 299
hypoglycaemic episodes | 3 | 7 | 3 | 5

25. Secondary Outcome: Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Percentage of subjects with treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes. A treatment emergent hypoglycaemic episode was defined as an episode with onset in the 'on-treatment' period (information collected while subjects were considered as exposed to trial product). This corresponded to information collected until the follow-up (5 weeks after the last treatment including a visit window of +7 days). Severe or BG-confirmed symptomatic hypoglycaemia was defined as an episode that was severe according to the American Diabetes Association classification or BG-confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: 40 weeks + follow-up of 5 weeks
Population: as for outcome 23
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 299
percentage of subjects | 0.7 | 1.7 | 1.0 | 1.7

26. Secondary Outcome: Change in Amylase
Description: as for outcome 9
Time Frame: Week 0, week 40
Population: Analysis was based on safety analysis set. Number of participants analysed=number of participants with available data for amylase.
Measure: Geometric Least Squares Mean (Standard Error); unit: ratio to baseline
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 295 | 296 | 292 | 294
ratio to baseline | 1.17 (0.02) | 1.22 (0.02) | 1.16 (0.02) | 1.20 (0.02)

27. Secondary Outcome: Change in Lipase
Description: as for outcome 9
Time Frame: Week 0, week 40
Population: Analysis was based on safety analysis set. Number of participants analysed=number of participants with available data for lipase.
Measure: Geometric Least Squares Mean (Standard Error); unit: ratio to baseline
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 295 | 296 | 291 | 293
ratio to baseline | 1.22 (0.04) | 1.32 (0.04) | 1.23 (0.04) | 1.29 (0.04)

28. Secondary Outcome: Change in Pulse Rate
Description: as for outcome 13
Time Frame: Week 0, week 40
Population: Analysis was based on safety analysis set.
Measure: Least Squares Mean (Standard Error); unit: beats/min
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 301 | 300 | 299 | 299
beats/min | 2.09 (0.51) | 3.96 (0.51) | 1.56 (0.49) | 2.42 (0.50)

ADVERSE EVENTS:
Time Frame: Baseline (week 0) to week 40 + follow up of 5 weeks (including a visit window of +7 days)
Description: A TEAE was defined as an AE with onset in the 'on-treatment' period (information collected while subjects were considered as exposed to trial product). This corresponded to information collected from first administration of trial product until the follow-up (5 weeks after the last treatment including a visit window of +7 days)
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Dulaglutide 0.75 mg | Dulaglutide 1.5 mg
All-Cause Mortality (participants affected / at risk) | 0/301 | 1/300 | 2/299 | 2/299
Serious Adverse Events (participants affected / at risk) | 17/301 | 23/300 | 24/299 | 22/299
Other Adverse Events (participants affected / at risk) | 132/301 | 134/300 | 106/299 | 139/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=301) | Semaglutide 1.0 mg (N=300) | Dulaglutide 0.75 mg (N=299) | Dulaglutide 1.5 mg (N=299)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardioversion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drowning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HIV infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orchidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatolithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=301) | Semaglutide 1.0 mg (N=300) | Dulaglutide 0.75 mg (N=299) | Dulaglutide 1.5 mg (N=299)
Constipation (Gastrointestinal disorders) | 16 (18) | 14 (14) | 10 (10) | 15 (18)
Decreased appetite (Metabolism and nutrition disorders) | 25 (26) | 27 (27) | 9 (12) | 31 (36)
Diarrhoea (Gastrointestinal disorders) | 43 (79) | 41 (96) | 23 (42) | 53 (75)
Headache (Nervous system disorders) | 25 (35) | 22 (30) | 12 (20) | 19 (30)
Lipase increased (Investigations) | 19 (23) | 17 (17) | 16 (17) | 17 (20)
Nasopharyngitis (Infections and infestations) | 15 (16) | 14 (16) | 17 (20) | 20 (24)
Nausea (Gastrointestinal disorders) | 67 (144) | 63 (192) | 39 (66) | 60 (108)
Upper respiratory tract infection (Infections and infestations) | 13 (18) | 10 (11) | 21 (26) | 16 (21)
Vomiting (Gastrointestinal disorders) | 30 (50) | 31 (48) | 12 (16) | 29 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT02648204/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT02648204/SAP_001.pdf